CLINICAL TRIAL: NCT00902304
Title: A Phase IV Clinical Trial of Intensified Blood Pressure Management in Primary Care Using Valsartan Alone and as Combination Anti-Hypertensive Therapy
Brief Title: Valsartan Intensified Primary Care Reduction of Blood Pressure Study
Acronym: VIPER-BP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489AAU01
Record Dates: First submitted 2009-04-28; First posted 2009-05-15 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: Hypertension; valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Active Comparator): Physicians applied their usual pattern of patient visits and treatment strategies to achieve individualized blood pressure target
  Interventions: Drug: Usual care
- Monotherapy (initial monotherapy arm) (Experimental): Physicians utilized valsartan 160mg per day for 6 weeks, followed by (if required) dose titrations every 4 weeks thereafter until week 14 (valsartan 320mg per day, then valsartan 320mg plus hydrochlorothiazide (HCTZ) 12.5mg per day, then valsartan 320mg plus HCTZ 25mg per day (maximal dose)). For patients not at blood pressure target at week 18, physicians were requested to consider triple or alternative therapy at their own discretion for the remainder of the study.
  Interventions: Drug: Valsartan and hydrochlorothiazide (HCTZ) - monotherapy; Drug: Valsartan
- Combination (initial combination therapy arm) (Experimental): Physicians initially utilized single tablet combination products of either valsartan plus hydrochlorothiazide (HCTZ) or valsartan plus amlodipine for an initial 6 weeks of therapy (based on the treating physician's preference), with dose titrations (if required) every 4 weeks thereafter until week 10. The maximum dose for the HCTZ combination was valsartan 160mg plus HCTZ 25mg per day. The maximum dose for the amlodipine combination was valsartan 160mg plus amlodipine 10mg per day. For patients who were not at blood pressure target at week 14, physicians were requested to consider triple or alternative therapy at their own discretion for the remainder of the study.
  Interventions: Drug: Valsartan and amlodipine; Drug: Valsartan and hydrochlorothiazide (HCTZ) - combination arm

INTERVENTIONS:
Drug: Valsartan and hydrochlorothiazide (HCTZ) - monotherapy — Monotherapy arm - if monotherapy valsartan 320mg per day orally was not sufficient, then could add HCTZ up to 25 mg per day orally
  Arms: Monotherapy (initial monotherapy arm)
Drug: Valsartan and amlodipine — From valsartan 80mg/amlodipine 5mg per day to valsartan 160mg/amlodipine 10mg per day orally
  Arms: Combination (initial combination therapy arm)
Drug: Usual care — As directed by investigator
  Arms: Usual care
Drug: Valsartan — Valsartan 160mg per day to 320mg per day orally
  Arms: Monotherapy (initial monotherapy arm)
Drug: Valsartan and hydrochlorothiazide (HCTZ) - combination arm — Combination arm - from valsartan 80mg/hydrochlorothiazide 12.5mg per day to valsartan 160mg/hydrochlorothiazide 25mg per day orally
  Arms: Combination (initial combination therapy arm)

SUMMARY:
This study will assess the efficacy of an intensive blood pressure management strategy compared to usual care in a primary care (general practice) setting.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or currently treated hypertensive patients who have not attained their blood pressure target and require active pharmacological treatment as recommended by the local guidelines as judged by the general practitioner

Exclusion Criteria:

* significantly elevated blood pressure (severe hypertension)
* requiring 3 or more antihypertensive drugs
* severe kidney disease or dialyses
* clinical diagnosis requiring concomitant therapy with antihypertensive treatment that would be outside the therapies allowed under study protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2337 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Australia (2):
  - Professor Garry Jennings-Co Principal Investigator, Melbourne
  - Professor Simon Stewart-Principal Investigator, Melbourne

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2337 patients were enrolled. 2185 received study medication during the 4 week run-in period. 1562 patients were randomized.
Period: Overall Study
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Started | 524 | 360 | 678
Completed | 466 | 289 | 568
Not Completed | 58 | 71 | 110
Not completed — Adverse Event | 4 | 10 | 25
Not completed — Investigator discretion | 3 | 5 | 13
Not completed — Lost to Follow-up | 7 | 7 | 7
Not completed — Protocol Violation | 9 | 18 | 20
Not completed — Withdrawal by Subject | 32 | 22 | 43
Not completed — includes pregnancy | 3 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm) | Total
Number analyzed (Participants) | 524 | 360 | 678 | 1562
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 59 (12) | 59 (12) | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 138 | 260 | 599
  Male | 323 | 222 | 418 | 963

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have Achieved Their Pre-specified (Individualized National Heart Foundation of Australia Criteria) Blood Pressure (BP) Target
Description: BP target groups were: <= 125/75mmHg, <= 130/80mmHg and <= 140/90mmHg. The BP target was based on the patient's clinical risk profile as specified by National Heart Foundation of Australia guidelines.
Time Frame: 26 weeks
Population: Intent-to-treat (ITT) - ITT population consisted of all subjects randomized to a study intervention arm and who commenced study management and/or treatment and who had at least one recorded BP post randomization. Last Observation Carried Forward (LOCF) imputation technique is used for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 504 | 339 | 649
percentage of participants | 27.4 | 33.0 | 37.9

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure
Description: The visit window was from 22 to 36 weeks. If more than one blood pressure measure was available within the specified window, then the one closest to the scheduled visit was used for analysis. If no measure was available within this window, then the last recorded BP post-randomization was used for the endpoint. Analysis of covariance model was used with the factors: baseline blood pressure, treatment and blood pressure target group at randomization.
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 504 | 339 | 649
mmHg | -10 [-11.3 to -8.8] | -11.6 [-13.1 to -10.0] | -14.4 [-15.5 to -13.2]

3. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 504 | 339 | 649
mmHg | -5.45 [-6.2 to -4.7] | -6.9 [-7.9 to -5.9] | -8.29 [-9.0 to -7.6]

4. Secondary Outcome: Change in Absolute Cardiovascular Risk Score
Description: The absolute cardiovascular risk assessment uses the Framingham Risk Equation to predict risk of a cardiovascular event over the next 5 years. A score of <10% is a low risk, 10 to 15% is a moderate risk, and >15% is a high risk.
  A decrease indicates improvement.
Time Frame: Baseline and 26 weeks
Population: Intent-to-treat (ITT) - ITT population consisted of all subjects randomized to a study intervention arm and who commenced study management and/or treatment and who had at least one recorded BP post randomization. Only patients with measurements at both baseline and week 26 were included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage risk score change
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 397 | 252 | 492
percentage risk score change | -2.6 (4.5) | -3.3 (4.6) | -3.9 (4.5)

5. Secondary Outcome: Number of Patients With at Least One Adverse Events Attributable to Anti-hypertensive Therapy
Description: The rate of all adverse events by preferred terms as determined by the General Practice investigators to be related to study intervention therapy was reported. Percentage of adverse events was calculated based on the number of participants analyzed. 41 adverse events were not reported as inadequate information was supplied to allow determination of drug treatment at onset.
Time Frame: 26 weeks
Population: Safety analysis - consisted of all subjects randomized to a study intervention arm and who commenced study management and/or treatment.
Measure: Number; unit: participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 524 | 360 | 678
participants | 70 | 70 | 169

6. Secondary Outcome: Number of 'Early Responder' Patients Who Achieve Individualized Blood Pressure Control After 1 or 2 Adjustments
Description: A comparison of the early responders was made based on the blood pressure measurements taken at the week 6 visit window according to gender and guideline targets. The guideline targets were: patients with renal impairment: 125/75 mmHg; patients with end-organ damage/cardiovascular disease: 130/80 mmHg; others: 140/90 mmHg.
Time Frame: 26 weeks
Population: Intent-to-treat (ITT) - ITT population consisted of all subjects randomized to a study intervention arm and who commenced study management and/or treatment and who had at least one recorded BP post randomization.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 524 | 360 | 678
Participants
  Male patients with a target of <125/75 mmHg | 3 | 3 | 6
  Male patients with a target of <130/80 mmHg | 27 | 14 | 34
  Male patients with a target of <140/90 mmHg | 31 | 22 | 48
  Female patients with a target of <125/75 mmHg | 2 | 2 | 2
  Female patients with a target of <130/80 mmHg | 16 | 5 | 34
  Female patients with a target of <140/90 mmHg | 18 | 11 | 42

7. Secondary Outcome: Change in the EQ-5D Score
Description: The EQ-5D total indexed score (AUS) measures self-reported quality of life with the following 5 dimensions: mobility (range 1,2,3), self-care (range 1,2,3), usual activity (range 1,2,3), pain/discomfort (range 1,2,3) and anxiety/depression (range 1,2,3), where a 1 indicates no problems, a 2 indicates moderate problems, and a 3 indicates severe problems. The range of possible utility scores are between -0.217 (derived from worse responses from all 5 dimensions with severe problems ie 3,3,3,3,3) and 1.000 (no problems for all 5 dimensions) for each dimension. An increase in EQ-5D indexed score (AUS) indicates improvement.
Time Frame: Baseline and 26 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: change in EQ-5D score
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 406 | 264 | 511
change in EQ-5D score | -0.007 [-0.022 to 0.008] | 0.017 [-0.001 to 0.036] | 0.011 [-0.003 to 0.024]

8. Secondary Outcome: Number of Patients With Depression
Description: Patients with depression refers to potential depressive symptoms, not clinically diagnosed depression. The 2 question Arrol screening tool was used to determine if the patient had potential depressive symptoms. The 2 questions are: During the last month have you often been bothered by feeling down, depressed or hopeless? During the past month have you often been bothered by little interest or pleasure in doing things? The presence of potential depressive symptoms was determined by a 'yes' answer to either of these questions.
Time Frame: Baseline and week 26
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 458 | 285 | 547
participants
  Baseline | 154 | 96 | 185
  Week 26 | 129 | 78 | 151

9. Secondary Outcome: Change in Center for Epidemiologic Studies Depression (CES-D) Score From Baseline to Week 26
Description: The CES-D score was from 0 to 30, with a higher score indicating a higher level of depression.
  The categories for the score are: 0 to 9 suggests no depression; 10 to 15 suggests mild depression; 16 to 24 suggests moderate depression; 24 or above suggests severe depression.
Time Frame: Baseline and week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: change in CES-D score
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 88 | 49 | 93
change in CES-D score | 1.03 (9.24) | -1.12 (10.95) | 1.19 (11.09)

10. Secondary Outcome: Participants With End Organ Disease at Baseline and Week 26
Description: A patient was considered to have end organ damage with either of the following: 1) proteinuria (dipstick = 1+ or more or protein/creatinine ratio > 30mg/mol or 24h urine protein > 0.3g); 2) no proteinuria, but presence of microalbuminuria (urine albumin/creatinine ratio 3.6 to 25mg/mol(male) or 3.6 to 35mg/mol (female) detected; 3) no proteinuria or microalbuminuria, but presence of macroalbuminuria (urine albumin/creatinine ratio > 25mg/mol(male) or >35mg/mol (female) detected OR 4) ECG evidence of LVH (Sokolow-Lyon voltage criteria values >= 38mm).
  Baseline potential for end organ damage was calculated in all 1562 randomised patients based on the criteria outlined above. If no investigation/data available, assumed no end-organ damage.
  It is important to note that given the limited number of ECGs at 26 weeks, between group comparisons should be limited to the two time points (baseline and 26 weeks).
Time Frame: Baseline and week 26
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 524 | 360 | 678
participants
  Baseline | 226 | 146 | 315
  Week 26 (N = 433, 277, 536) | 157 | 88 | 177

11. Secondary Outcome: Change in Self-care Behavior Score From Baseline to Week 26
Description: A modified self-care behavior tool (questionnaire) was used to calculate 2 domain scales: maintenance and confidence. Each domain has a standardized score between 0 and 100. Self-care is best represented by maintenance. Confidence is an important process that moderates the relationship between self-care and outcomes. Higher index score suggests better self-care. A score of 70 or greater can be used as the cut-point to judge self-care adequacy.
Time Frame: Baseline and week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Change in score
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 426 | 273 | 523
Change in score
  Maintenance score | 2.59 (13.56) | 2.27 (12.56) | 3.17 (12.38)
  Confidence score (N = 422, 269, 520) | 0.93 (21.04) | -0.72 (20.04) | -0.71 (20.16)

12. Secondary Outcome: Rate of Treatment Compliance
Description: The rate of compliance was planned to be estimated from the quantity of unused medication returned at each scheduled visit over the entire follow-up period. Rate of compliance = (tablets supplied - tablets returned)/(tablets for 100% compliance).
Time Frame: 26 weeks
Population: This data will not be analyzed due to the poor quality of the data.
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Patients With Major Clinical Endpoints
Description: Major clinical endpoints measured were all-cause mortality and fatal and non-fatal cardiovascular events (e.g. acute myocardial infarction, stroke and heart failure).
Time Frame: 26 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Number analyzed (Participants) | 524 | 360 | 678
participants
  All-cause mortality | 0 | 1 | 0
  Non-fatal cardiovascular events | 15 | 6 | 13

ADVERSE EVENTS:
Groups:
- Pre-randomization: Pre-randomization
Arm/Group | Pre-randomization | Usual Care | Monotherapy (Initial Monotherapy Arm) | Combination (Initial Combination Therapy Arm)
Serious Adverse Events (participants affected / at risk) | 27/2185 | 24/524 | 15/360 | 22/678
Other Adverse Events (participants affected / at risk) | 95/2185 | 47/524 | 36/360 | 105/678
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-randomization (N=2185) | Usual Care (N=524) | Monotherapy (Initial Monotherapy Arm) (N=360) | Combination (Initial Combination Therapy Arm) (N=678)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 3 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Chest discomfort (Cardiac disorders) | 0 | 2 | 0 | 0
Chest pain (Cardiac disorders) | 2 | 1 | 1 | 5
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Dizziness (Cardiac disorders) | 1 | 1 | 0 | 1
Dyspnoea (Cardiac disorders) | 0 | 3 | 1 | 4
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Syncope (Cardiac disorders) | 1 | 2 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enlarged uvula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Pseudocyst (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Biopsy prostate (Investigations) | 1 | 0 | 0 | 0
Blood test abnormal (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Vitamin B12 increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cystosarcoma phyllodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Exertional headache (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional drug misuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Arthroscopic surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-randomization (N=2185) | Usual Care (N=524) | Monotherapy (Initial Monotherapy Arm) (N=360) | Combination (Initial Combination Therapy Arm) (N=678)
Dizziness (Cardiac disorders) | 77 | 23 | 28 | 42
Oedema peripheral (General disorders) | 20 | 27 | 9 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.